CLINICAL TRIAL: NCT06937099
Title: A Phase 3b, Randomized, Multicenter, Controlled Study of Mirikizumab and Placebo or Mirikizumab Concomitantly Administered With Tirzepatide in Adult Participants With Moderately to Severely Active Crohn's Disease and Obesity or Overweight
Brief Title: Mirikizumab and Tirzepatide Administered in Adult Participants With Moderately to Severely Active Crohn's Disease and Obesity or Overweight
Acronym: COMMIT-CD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27281; 2024-520210-21-00 (EU CTIS Number); I6T-MC-AMCE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-18; First posted 2025-04-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease; Obesity or Overweight
MeSH Terms: conditions — Crohn Disease; Obesity; Overweight | interventions — mirikizumab; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Mirikizumab will be open label, tirzepatide and placebo to match will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mirikizumab + Tirzepatide (Experimental): Mirikizumab administered intravenously (IV) then Mirikizumab administered subcutaneously (SC).
  Tirzepatide administered SC.
  Interventions: Drug: Mirikizumab; Drug: Tirzepatide
- Mirikizumab + Placebo (Experimental): Mirikizumab administered IV then Mirikizumab administered SC. Placebo administered SC.
  Interventions: Drug: Mirikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Mirikizumab — Administered IV
  Other Names: LY3074828
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Mirikizumab + Tirzepatide
Drug: Placebo — Administered SC
  Arms: Mirikizumab + Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of mirikizumab and placebo compared with mirikizumab and concomitantly administered tirzepatide in adult participants with moderately to severely active CD and obesity, or overweight.

The maximum duration of this study is up to 61 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of Crohn's disease (CD) or perianal fistulizing CD
* Have obesity body mass index 30 kilograms per meter squared (BMI ≥30 kg/m²), or overweight (BMI ≥27 kg/m2 to <30 kg/m²) and in the presence of at least 1 weight-related comorbid conditions:

  * hypertension
  * Type 2 diabetes mellitus (T2DM)
  * dyslipidemia
  * obstructive sleep apnea, or
  * cardiovascular disease.
* Have moderately to severely active CD defined by a CDAI score of at least 220 at baseline.
* Have a centrally read Simple Endoscopic Score for Crohn's Disease (SES-CD) score ≥6 for patients with ileal-colonic or ≥4 for patients with isolated ileal disease within 21 days before the first dose of study treatment.
* Participants with a history of CD for ≥8 years involving only or predominantly the colon must have documented negative results for colorectal dysplasia and cancer within 1 year prior to baseline.
* Demonstrated inadequate response, loss of response or intolerance to at least one protocol-specified conventional or advanced CD therapy

Exclusion Criteria:

* Have a current diagnosis of Ulcerative Colitis (UC), inflammatory bowel disease-unclassified (formerly known as indeterminate colitis), or primary sclerosing cholangitis.
* Have more than 2 missing segments of the following 5 segments: terminal ileum, ·right colon, transverse colon, ·left colon, and rectum.
* Currently have or are suspected to have an abscess.
* Have a stoma, ileoanal pouch, or ostomy.
* Have a history of more than 3 small bowel resections, total resection of small bowel greater than 100 centimeters (cm), diagnosis of short bowel syndrome, or any intestinal or non-intestinal intra-abdominal surgery within 3 months of baseline.
* Have a diagnosis of Type 1 Diabetes Mellitus (T1DM) or have insulin-treated T2DM.
* Have a history of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to screening.
* Have had more than 5% body weight change in the past 3 months
* Have a current or recent acute, active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Simultaneously Achieve Clinical Remission by Crohn's Disease Activity Index (CDAI), Endoscopic Remission, and at least 10% Weight Reduction | Week 52
  Percentage of participants who simultaneously achieve clinical remission by CDAI, endoscopic remission and at least 10% weight reduction.

SECONDARY OUTCOMES:
Percentage of Participants Who Simultaneously Achieve Clinical Remission by CDAI and Endoscopic Remission | Week 24, 52
  Percentage of participants who simultaneously achieve clinical remission by CDAI and endoscopic remission.
Percentage of Participants Who Achieved Maintenance of Clinical Remission by CDAI | Week 52
  Percentage of participants who achieve maintenance of clinical remission by CDAI.
Percentage of Participants Who Achieved Maintenance of Endoscopic Remission | Week 52
  Percentage of participants who achieve maintenance of endoscopic remission.
Percentage of Participants Who Achieve Corticosteroid-free Clinical Remission by CDAI Among Participants Who Used Corticosteroids at Baseline | Week 52
  Percentage of participants who achieve corticosteroid-free clinical remission by CDAI among participants who used corticosteroids at baseline.
Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) | Baseline, Week 52
  Change from baseline in inflammatory bowel disease questionnaire (IBDQ).
Percentage of Participants Who Achieve at Least a 10% Reduction in Body Weight | Week 52
  Percentage of participants who achieve at least a 10% reduction in body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (185):
- United States (35):
  - Digestive Health Specialists, Dothan, Alabama
  - Smart Cures Clinical Research, Anaheim, California
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - United Medical Doctors - Los Alamitos, Los Alamitos, California
  - California Medical Research Associates, Northridge, California
  - Research Associates of South Florida - Miami - Southwest 8th Street, Miami, Florida
  - Gastro Health Research - Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Gastro Health Research - Pensacola, Pensacola, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Gastroenterology Health Partners, New Albany, Indiana
  - Gastroenterology Health Partners, Louisville, Kentucky
  - Care Access - New Iberia, New Iberia, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Capital Digestive Care - Chevy Chase, Chevy Chase, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Gastroenterology Associates, New York, New York
  - Care Access - Yonkers, Yonkers, New York
  - Coastal Research Institute - Fayetteville, Fayetteville, North Carolina
  - Gastro Intestinal Research Institute of Northern Ohio, LLC, Westlake, Ohio
  - Thomas Jefferson University - Medicine/GI and Hepatology, Philadelphia, Pennsylvania
  - University Gastroenterology - Providence - West River Street, Providence, Rhode Island
  - Gastroenterology Associates - Patewood, Greenville, South Carolina
  - Gastroenterology Center Of The Midsouth, Cordova, Tennessee
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Southern Star Research Institute, San Antonio, Texas
  - Tyler Research Institute, Tyler, Texas
  - Washington Gastroenterology - Tacoma, Tacoma, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Belgium (6):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
  - Clinical Chc Montlégia, Liège
- Brazil (15):
  - NewData Clinical Research - Aracaju, Aracaju
  - L2IP - Instituto de Pesquisas Clínicas, Brasília
  - Loema Instituto de Pesquisa Clinica, Campinas
  - Fundação Universidade de Caxias do Sul (FUCS), Caxias do Sul
  - Centro Digestivo de Curitiba, Curitiba
  - Galileo Medical Research, Juiz de Fora
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - CLIAGEN Clínica de Atenção em Gastroenterologia, Especialidades e Nutrição, Salvador
  - Pesquisare Saude, Santo André
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Clínica Hepatogastro JK, São Paulo
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Bulgaria (3):
  - University Hospital "St. Ivan Rilski", Gorna Oryahovitsa
  - Multiprofile Hospital for Active Treatment "Knyaginya Klementina" - Sofia EAD, Sofia
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna-ISUL" EAD, Sofia
- Canada (6):
  - Gastroenterology and internal medicine research institute, Edmonton
  - Victoria Hospital & Children's Hospital - London Health Sciences Centre, London
  - London Digestive Disease Institute, London
  - Clinique IMD, Montreal
  - Vancouver General Hospital, Vancouver
  - (G.I.R.I.) GI Research Institute Foundation, Vancouver
- Czechia (6):
  - SurGal Clinic, Brno
  - Gastroenterologie, Hradec Králové
  - EndoArt, Ostrava
  - ResTrial GastroEndo s.r.o, Prague
  - ISCARE klinické centrum, Prague
  - Masarykova Nemocnice V Usti Nad Labem, Ústí nad Labem
- Denmark (5):
  - Aalborg Universitetshospital, Syd, Aalborg
  - Aarhus Universitetshospital, Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Copenhagen
  - Vejle Sygehus, Vejle
- France (11):
  - Clinique des Cèdres, Échirolles
  - CHD Vendee, La Roche-sur-Yon
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Chu Saint Eloi, Montpellier
  - Centres Médico Chirurgicaux - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Hôpital Saint Antoine, Paris
  - CHU Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord, Saint-Priest-en-Jarez
  - CHU Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (6):
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Praxiszentrum für Gastroenterologie, Grevenbroich
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Eugastro GmbH, Leipzig
  - Klinikum Ernst von Bergmann, Potsdam
- Greece (5):
  - Evangelismos General Hospital of Athens, Athens
  - Thoracic General Hospital of Athens "I Sotiria", Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - CLINFAN Szolgáltató Kft, Szekszárd
- Israel (8):
  - Assuta Ashdod Medical Center, Ashdod
  - Rambam Health Care Campus, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (10):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Ospedale Specializzato in Gastroenterologia "Saverio de Bellis", Castellana Grotte
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedale - Università Padova, Padua
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Di Circolo, Rho
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Humanitas, Rozzano
- Mexico (16):
  - San Peregrino Unidad de Investigación, Aguascalientes
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Boca Clinical Trials Mexico S.C., Guadajalara
  - Centro de Investigación Clínica y Medicina Traslacional (CIMeT), Guadalajara
  - Hospital General de Occidente, Guadalajara
  - Health Pharma Querétaro, Juriquilla
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Medical Care and Research SA de CV, Mérida
  - Servicios de Oncología Médica Integral - Monterrey, Monterrey
  - Centro de Investigacion Clinica Chapultepec, Morelia
  - Boca Clinical Trials Mexico SC, Puebla City
  - Clinical Research Institute S.C., Tlalnepantla
  - FAICIC S. de R.L. de C.V., Veracruz
- Netherlands (5):
  - Amsterdam UMC, locatie VUmc, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (12):
  - Medrise Sp. z o.o., Lublin
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - IRMED, Piotrkow Trybunalski
  - Twoja Przychodnia PCM, Poznan
  - Uniwersyteckie Centrum Stomatologii i Medycyny Specjalistycznej, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Twoja Przychodnia SCM, Szczecin
  - NZOZ GynCentrum - Oddział Warszawa, Warsaw
  - Vivamed Sp. z o.o., Warsaw
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw
  - Melita Medical, Wroclaw
  - ETG Zamość, Zamość
- CMRC Headlands, LLC, San Juan, Puerto Rico
- Romania (6):
  - Spitalul Județean de Urgență Bacău, Bacau
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Universitar de Urgență București, Bucharest
  - Constanta County Emergency Clinical Hospital Sf.Ap.Andrei, Constanța
  - Spitalul Clinic Județean de Urgență, Craiova
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - ENDOMED, Košice
  - Gastro LM, Prešov
- Spain (10):
  - Centro Médico Teknon, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Arquitecto Marcide, Ferrol
  - Hospital de Cabueñes, Gijón
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (9):
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Uludag Universitesi, Bursa
  - Eskisehir Osmangazi University, Eskişehir
  - Mustafa Kemal Universitesi, Hatay
  - Bezmialem Vakf Üniversitesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - Kocaeli University Medical Faculty Hospital, İzmit
  - Mersin University, Mersin
  - Antalya Egitim ve Arastırma Hastanesi, Muratpaşa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/600156